CLINICAL TRIAL: NCT00054691
Title: A Phase II Study of ZD1839 (Iressa), Epidermal Growth Factor Receptor (EGFR) Tyrosine Kinase Inhibitor, in Treatment of Recurrent or Metastatic Squamous Cell Carcinoma of the Skin
Brief Title: ZD1839 (Iressa) for Recurrent or Metastatic Squamous Cell Carcinoma of the Skin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID02-282
Record Dates: First submitted 2003-02-06; First posted 2003-02-07 (Estimated); Results first posted 2015-02-12 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-02

CONDITIONS: Skin Cancer
Keywords: Skin Cancer; Squamous Cell Carcinoma of the Skin; Gefitinib; ZD1839; Iressa; Epidermal Growth Factor Receptor; EGFR
MeSH Terms: conditions — Skin Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iressa (ZD1839) (Experimental): Iressa (ZD1839) 250 mg by mouth daily.
  Interventions: Drug: Iressa

INTERVENTIONS:
Drug: Iressa — 250 mg by mouth daily
  Other Names: ZD1839; Gefitinib

SUMMARY:
The goal of this clinical research study is to learn if the drug ZD1839 (Iressa) can shrink or slow the growth of cancer in participants with recurrent and/or metastatic squamous cell cancer (SCC) of the skin. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
ZD1839 is a new drug that may slow or stop cell growth in humans.

Epidermal growth factor receptor (EGFR) may be involved in certain types of cancer, including squamous cell carcinoma of the skin. When EGFR is stimulated, a series of chemical reactions starts that results in a tumor being "told" to grow. ZD1839 tries to stop these reactions by blocking EGFR. This may stop tumors from growing.

In this study, participants will take ZD1839 by mouth daily. Once the treatment has started, participants will return to the clinic before every treatment cycle (every 4 weeks) for the first 4 months then every 8 weeks thereafter. At these visits, participants will have a physical exam and blood tests will be performed. About 2-4 teaspoons of blood will be drawn at each visit. The doctor will also check on how participants are tolerating ZD1839 (side effects). Every 8 weeks, participants will have their tumor evaluated by radiographic scans. This may include either a CT or MRI and a chest X-ray.

During treatment, participants should not take any other medication, including non-prescription drugs such as aspirin or herbal products without the approval of their doctor.

Participants will continue taking the trial drug until the tumor grows, a severe side effect occurs, they withdraw consent, or the study is closed. The study will be closed 12 months after the last participant is enrolled.

This is an investigational study. The FDA has approved ZD1839 for the treatment of advanced lung cancer, but the FDA has authorized ZD1839 for research only in the treatment of skin cancer. About 40 participants will take part in this study. All will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent.
2. Pathologically confirmed locoregional recurrence and/or metastatic SCC of the skin not amenable to curative therapy (i.e., surgery or radiation).
3. Evaluable and/or measurable disease. (Based on Union for International Cancer Control (UICC)/World Health Organization (WHO) Criteria)
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
5. Adequate hematologic function as defined by an absolute neutrophil count >= 1,500/mm3, a platelet count >= 100,000/mm3, a white blood count (WBC) >= 3,000/ mm3, and a hemoglobin level of >= 9 g/dl.
6. Up to one prior chemotherapy regimen.
7. At least a 2-week recovery from prior therapy toxicity.
8. Age 18 years or older.
9. Disease free from a previously treated malignancy, other than the disease under study, for greater than 3 years. Patients with a history of a previous basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix, completely resected breast cancer will not be excluded.
10. Women of childbearing potential and men must be willing to practice acceptable methods of birth control to prevent pregnancy.

Exclusion Criteria:

1. Prior ZD1839 or other Epidermal growth factor receptor (EGFR) inhibiting agents.
2. Other co-existing malignancies or malignancies diagnosed within the last 3 years with the exception of basal cell carcinoma or cervical cancer in situ.
3. Any unresolved chronic toxicity greater then Common Terminology Criteria (CTC) grade 2 from previous anticancer therapy.
4. Incomplete healing from previous oncologic or other major surgery.
5. Concomitant use of phenytoin, carbamazepine, barbiturates, rifampicin, St John's Wort. Patients taking anticoagulants must have coagulation parameters followed (i.e., Prothrombin time (PT) or Partial thromboplastin time (PTT)).
6. Absolute neutrophil count (ANC) less than 1,500/mm**3 or platelets less than 100,000/mm**3.
7. Serum bilirubin greater than 1.25 times the upper limit of reference range (ULRR).
8. In the opinion of the investigator, any evidence of severe or uncontrolled systemic disease, (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease).
9. Alanine amino transferase (ALT) or aspartate amino transferase (AST) greater than 2.5 times the ULRR if no demonstrable liver metastases or greater than 5 times the Upper Limit of the Reference Range (ULRR) in the presence of liver metastases.
10. Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the trial.
11. Pregnancy or breast feeding (women of child-bearing potential)
12. The patient has an uncontrolled seizure disorder or active neurological disease.
13. The patient has received any non-approved or investigational agent(s) within 30 days before Day 1 of study treatment.
14. Known, severe hypersensitivity to ZD1839 or any of the excipients of this product.
15. Any evidence of clinically active Interstitial Lung Disease (ILD) (patients with chronic, stable radiographic changes who are asymptomatic need not be excluded).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie S. Glisson, MD, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: July 2004 to September 2007. All participants recruited at The University of Texas MD Anderson Cancer Center.
Groups:
- Iressa (ZD1839): 250 mg by mouth daily (1 course = 4 weeks), 6 courses of treatment.
Period: Overall Study
Arm/Group | Iressa (ZD1839)
Started | 40
Completed | 37
Not Completed | 3
Not completed — Unmeasurable Disease | 2
Not completed — Noncompliant | 1

BASELINE CHARACTERISTICS:
Population: Out of 40 participants, 2 participants had unmeasurable disease and 1 participant was noncompliant.
Arm/Group | Iressa (ZD1839)
Number analyzed (Participants) | 40
Age, Customized [Median (Full Range); unit: years] | 67 [37 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 30
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response (Partial Response, Stable Disease and Progressive Disease)
Description: Responses were assessed according to the Union Internationale Contre le Cancer (UICC) / World Health Organization (WHO) criteria. Objective response (measurable response) defined as: Partial response (PR): Applies only to participants with at least 1 measurable lesion; >/=50% decrease under baseline in sum of products of perpendicular diameters of all measurable lesions. Stable Disease (SD): No progression of evaluable disease and/or no new lesions. Progressive Disease (PD): 50% increase or an increase of 10 cm2 (whichever is smaller) in the sum of products of all measurable lesions overall smallest sum observed (over baseline if no decrease) using the same techniques as baseline, OR clear worsening of any evaluable disease.
Time Frame: Every 8 weeks till disease progression.
Population: Out of 40 participants, 2 participants had unmeasurable disease and 1 participant was noncompliant.
Measure: Number; unit: participants
Arm/Group | Iressa (ZD1839)
Number analyzed (Participants) | 37
participants
  Stable Disease | 14
  Partial Response | 4
  Progressive Disease | 19

2. Secondary Outcome: Duration of Response
Description: Response duration was defined as the time from initial response during therapy to progression of disease.
Time Frame: Every 8 weeks till disease progression.
Population: Out of 40 participants, 19 participants had progressive disease, 2 participants had unmeasurable disease and 1 participant was noncompliant.
Measure: Median (Full Range); unit: months
Arm/Group | Iressa (ZD1839)
Number analyzed (Participants) | 18
months | 24.8 [0.9 to 47.2]

ADVERSE EVENTS:
Time Frame: Reporting Period: November 2007 to September 2009.
Arm/Group | Iressa (ZD1839)
Serious Adverse Events (participants affected / at risk) | 17/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iressa (ZD1839) (N=40)
Pulmonary Embolism (Vascular disorders) | 3 (4)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Intestinal Ischaemia (Gastrointestinal disorders) | 1 (1)
Pseudotumor Cerebri (Musculoskeletal and connective tissue disorders) | 1 (1)
Severe Gastrointestinal Bleeding (Melena) (Gastrointestinal disorders) | 1 (1)
Pharyngeal Mucositis (Immune system disorders) | 1 (1)
Stomatitis (Immune system disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Leptomeningeal Metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Bone Marrow Depression (Blood and lymphatic system disorders) | 1 (1)
Deep Vein Thrombosis (Legs) (Vascular disorders) | 2 (2)
Ruptured Superior Vena Cava (Injury, poisoning and procedural complications) | 1 (1)
Chronic Pulmonary Thromboembolism (Vascular disorders) | 1 (1)
Hepatic Function Disorder (Hepatobiliary disorders) | 2 (2)
Blood Creatinine, Increased (Blood and lymphatic system disorders) | 1 (1)
Worsening Hypertension (Cardiac disorders) | 1 (1)
Worsening Renal Function (Renal and urinary disorders) | 1 (1)
Thrombosis of Goretex (Vascular disorders) | 1 (1)
Worsening of Migraine (General disorders) | 1 (1)
Interstitial Pneumonia (Infections and infestations) | 2 (2)
Odynophagia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Myeloid Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Weakness (General disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iressa (ZD1839) (N=40)
ACNE (Skin and subcutaneous tissue disorders) | 3 (3)
ALLERGIC RHINITIS (General disorders) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 (2)
ALT, SGPT (Hepatobiliary disorders) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 1 (1)
ANOREXIA (Psychiatric disorders) | 5 (5)
AST, SGOT (Hepatobiliary disorders) | 2 (2)
BUN INCREASE (Hepatobiliary disorders) | 3 (3)
CHEILITIS (Immune system disorders) | 2 (2)
CONSTIPATION (Gastrointestinal disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2)
CREATININE INCREASE (Hepatobiliary disorders) | 1 (1)
DEHYDRATION (General disorders) | 2 (2)
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1)
DERMATOLOGY/SKIN (Skin and subcutaneous tissue disorders) | 4 (4)
DIARRHEA (Gastrointestinal disorders) | 22 (22)
DIZZINESS (General disorders) | 2 (2)
DRY SKIN (Skin and subcutaneous tissue disorders) | 6 (6)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 4 (4)
EDEMA: HEAD AND NECK (Vascular disorders) | 1 (1)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 2 (2)
FATIGUE (General disorders) | 16 (16)
FEVER WITHOUT NEUTROPENIA (General disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
HEARTBURN (Gastrointestinal disorders) | 1 (1)
HEMOGLOBIN (Blood and lymphatic system disorders) | 1 (1)
PULMONARY HEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 2 (2)
HYPERGLYCEMIA (Endocrine disorders) | 1 (1)
HYPERKALEMIA (Blood and lymphatic system disorders) | 1 (1)
HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 3 (3)
HYPERURICEMIA (Hepatobiliary disorders) | 1 (1)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 6 (6)
INFECTION (Infections and infestations) | 3 (3)
INTERNATIONAL NORMALIZED RATIO (Blood and lymphatic system disorders) | 1 (1)
KERATITIS (Infections and infestations) | 1 (1)
LEUKOCYTES (Immune system disorders) | 1 (1)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1)
METABOLIC (Metabolism and nutrition disorders) | 1 (1)
MUCOSITIS (Immune system disorders) | 1 (1)
NAIL CHANGES (Skin and subcutaneous tissue disorders) | 2 (2)
NAUSEA (General disorders) | 5 (5)
OCULAR/VISUAL (Eye disorders) | 1 (1)
PAIN (General disorders) | 1 (1)
PAIN (ABDOMEN NOS) (Gastrointestinal disorders) | 1 (1)
PAIN (JOINT) (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN (ORAL CAVITY) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN (STOMACH) (Gastrointestinal disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 5 (5)
RASH ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 26 (26)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SYNCOPE (FAINTING) (Nervous system disorders) | 1 (1)
VERTIGO (Nervous system disorders) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
WATERY EYES (Eye disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No